CLINICAL TRIAL: NCT00615082
Title: Stress Reduction for Caregivers: A Randomized Controlled Pilot Study
Brief Title: The Balance Study Balancing Life and Reducing Stress For Those Providing Elder Care
Acronym: Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1R21AT003654-01A1 (NIH); R21AT003654-01A1 (NIH)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2011-09

CONDITIONS: Dementia; Caregivers; Stress
MeSH Terms: conditions — Dementia | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): Behavioral: Mindfulness-Based Stress Reduction
  Other Names:
  MBSR An 8-week course led by an experienced instructor in a group format of up to 15 people. Participants in the MBSR course learn mindfulness meditation techniques and simple yoga exercises such as stretching.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Caregiver Education & Social Support (Active Comparator): Behavioral: Caregiver Education & Social Support
  Other Names:
  CESS An 8-week course led by experienced instructors in a group format of up to 15 people. Participants in the CESS course learn about a variety of important issues related to elder care and receive social and emotional support in a group discussion format.
  Interventions: Behavioral: Caregiver Education & Social Support

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — An 8-week course led by an experienced instructor in a group format of up to 15 people. Participants in the MBSR course learn mindfulness meditation techniques and simple yoga exercises such as stretching.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Caregiver Education & Social Support — An 8-week course led by experienced instructors in a group format of up to 15 people. Participants in the CESS course learn about a variety of important issues related to elder care and receive social and emotional support in a group discussion format.
  Other Names: CESS
  Arms: Caregiver Education & Social Support

SUMMARY:
The primary goals of this exploratory/developmental (R21) study are to evaluate the feasibility and acceptability of a MBSR intervention for caregivers of patients with dementia, and to estimate the effectiveness of program outcomes on standardized measures of perceived stress, psychological distress and caregiver burden. We will randomize 60 caregivers 1:1 to participate in: 1.) an intervention arm consisting of a MBSR program that includes 8 weeks of group instruction in mindfulness meditation techniques followed by home practice, or 2.) an active control arm consisting of a standard 8 week Community Caregiver Education and Support (CESS) program.

DETAILED DESCRIPTION:
We anticipate that caregivers will be interested in participating in the intervention, be open to randomization, and have good rates of compliance with the program. It is also expected that MBSR program participants will evidence a trend toward better outcomes than CESS participants on primary outcome measures of perceived stress, psychological distress and perceived caregiver burden.

Substudy The purpose of this proposal is to add a physiologic outcome sub-study to the Balance project that will examine four biological markers correlated with stress in caregivers participating in the study intervention. The Balance Study is a recently funded NIH randomized controlled pilot study to evaluate the acceptability and feasibility of a Mindfulness-Based Stress Reduction (MBSR) intervention for caregivers of patients with dementia. Balance is randomizing caregivers (N=60) into equal numbers to participate in either an intervention arm consisting of a MBSR program that includes eight weeks of group instruction in mindfulness meditation techniques followed by home practice or an active control arm consisting of a standard eight week community Caregiver Education and Social Support (CESS) program. The specific aims of this study are to: 1) evaluate the feasibility of adding physiologic markers to the Balance Study; 2) examine changes over time in individual study participants on four biological markers correlated with stress including interleukin 6 (IL-6), D-dimer, DHEA-S and telomere length; and 3) to examine preliminary differences between MBSR and CESS groups on four biological markers. The addition of physiologic outcomes to the Balance Study presents an emerging opportunity to increase the competitiveness for our NIH R01 application.

ELIGIBILITY:
Inclusion Criteria:

* adult, 21 or older
* caregiver for a community dwelling patient with dementia
* English speaking
* literate - able to read course materials
* mentally intact with no history of mental illness
* reachable by phone
* able to attend weekly classes in the Bloomington area
* interested in either type of program (psycho-educational/mind-body intervention)
* willing to complete an informed consent process
* willing to be randomized and participate in one of two interventions
* experiencing significant stress (scale of 1-10 score of 5 or higher)

Exclusion Criteria:

* have previously participated in a community caregiver education and support group
* have previously completed formal training in other mind body practices such as meditation, yoga, or tai chi, or who are currently practicing
* are regularly practicing mindfulness meditation
* express uncertainty that they can attend the intervention on a regular basis
* not experiencing significant stress

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of conducting a trial comparing mindfulness-based stress reduction (MBSR) and community caregiver education and support (CESS) programs on stress reduction for caregivers of patients with dementia. | through study completion, an average of 1 year
  participants will complete surveys and consent to a blood draw at baseline, post intervention, and 6 months. They will complete a daily health behaviors calendar, and a subset will track their daily blood pressure.

SECONDARY OUTCOMES:
Estimate the effectiveness of a MBSR program compared to a standard CESS program for caregivers of persons with dementia. | through study completion, an average of 1 year
  participants will complete surveys and consent to a blood draw at baseline, post intervention, and 6 months. They will complete a daily health behaviors calendar, and a subset will track their daily blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whitebird, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States